CLINICAL TRIAL: NCT00488319
Title: A 6-Month, Open-Label, Single-Arm Safety Study of Flexibly Dosed Paliperidone Extended Release (1.5 - 12 mg/Day) in the Treatment of Adolescents (12 to 17 Years of Age) With Schizophrenia
Brief Title: Open-label Study of Flexible-dose Paliperidone ER (Extended Release) to Treat Adolescent Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012616; R076477PSZ3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2013-11

CONDITIONS: Schizophrenia; Schizophrenic Disorders; Psychotic Disorders; Dementia Praecox
Keywords: Schizophrenia; Adolescent; Paliperidone; Antipsychotic agents; Antipsychotic drugs; Psychosis.
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Paliperidone ER1.5 to 12 mg tablet once daily for 6 months
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — 1.5 to 12 mg tablet once daily for 6 months

SUMMARY:
The purpose of this open-label study is to evaluate the long-term (6-month) safety and tolerability of extended-release paliperidone, an atypical antipsychotic, given in flexible dosages to adolescents with schizophrenia.

DETAILED DESCRIPTION:
This is a 6-month, open-label study (the patient, investigator, and sponsor know the study drug and dosage being taken by the patient) of the safety and tolerability of flexible-dose (1.5 to 12mg per day), extended-release (ER) paliperidone in adolescents with a diagnosis of schizophrenia. Patients who have completed study R076477PSZ3001 or who discontinued from that study because of lack of efficacy but completed a minimum of 21 days of the study may enter this study. Patients may also enter this study directly without participating in R076477PSZ3001. This study consists of a 21-day screening and washout phase (to discontinue and "wash out" any medication not allowed in the study), an open-label treatment phase of up to 26 weeks during which all patients will take oral paliperidone ER every day, and a post-treatment phase consisting of a follow-up visit completed 1 week after a patient has received the final dose of paliperidone ER. The study, including the screening and posttreatment phase, will last approximately 30 weeks. Screening and washout may be conducted while a patient is either an inpatient or an outpatient. Safety will be assessed by laboratory measurements (chemistry, liver function tests, hematology, hormone, lipid assessments, prolactin [blinded], urinalysis, and urine drug screens); body weight, height, and waist circumference measurements; ECGs; and physical examinations (including Tanner staging). The Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson Angus Rating Scale (SAS) will be used to assess extrapyramidal symptoms (EPS) and dyskinesias. Adverse events will be monitored including psychiatric adverse events of interest (i.e., suicide and related phenomena, homicidal ideation, depressed mood, and worsening of psychosis) that may be associated with paliperidone ER in this population. The primary aim of this study is to evaluate the long-term (6-month) safety and tolerability of paliperidone ER in adolescents with schizophrenia. As exploratory secondary aims, the study will assess the effect of paliperidone ER on the long-term symptoms of schizophrenia as measured by the changes in the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scores, the global improvement in severity of illness as measured by the Clinical Global Impression-Severity (CGI-S) scale, the benefits in psychological, social, and school functioning as measured by the Children's Global Assessment Scale (CGAS), the changes in multiple domains of cognitive functioning measured by the modified Measurements and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) assessment battery, and the effect on sleep as measured by the sleep Visual Analog Scale (VAS). Patients begin the study at 6.0 mg/day of oral paliperidone ER. If a higher dosage is needed, the dosage will be increased (in increments of 3 mg/day not more frequently than once every 5 days) to 12 mg/day. If the 6.0 mg/day dosage is not well tolerated, the dosage may be decreased (not more frequently than once every 5 days) to 3.0 mg/day or 1.5 mg/day. Patients will be dosed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-IV criteria for schizophrenia, otherwise physically healthy
* Weight >=63.9 pounds (29 kg)
* Must not be a danger to self or others and must have family support available to be maintained as outpatients
* Responsible adult must be available to accompany the patient to the investigational site at each visit.

Exclusion Criteria:

* Meets the DSM-IV criteria for dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, or primary substance-induced psychotic disorder
* mild, moderate, or severe mental retardation
* History of substance dependence (including alcohol, but excluding nicotine and caffeine) according to the DSM-IV criteria in the 3 months before screening
* pregnancy (for females)
* History or presence of circumstances that may increase the risk of the occurrence of torsade de pointes or sudden death in association with the use of drugs that prolong the QTc interval.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (14):
  - Cerritos, California
  - San Diego, California
  - Santa Ana, California
  - Middletown, Connecticut
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Las Vegas, Nevada
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
- Antwerp, Belgium
- Sofia, Bulgaria
- Estonia (3):
  - Tallinn
  - Tartu
  - Viljandi
- Finland (2):
  - Hus
  - Kellokoski
- India (4):
  - Chennai
  - Hyderabad
  - Mangalore
  - Varanasi
- Poland (6):
  - Gdansk
  - Lódź
  - Poznan
  - Sosnowiec
  - Torun
  - Warsaw
- Bucharest, Romania
- Russia (11):
  - Ekaterinburg Na
  - Kazan'
  - Moscow
  - Moscow Russia
  - Nizhny Novgorod
  - Saint Petersburg
  - Saratov
  - Smolensk Region N/A
  - Stavropol Na
  - Tomsk Na
  - Yaroslavl
- South Korea (4):
  - Cheonan
  - Gyeonggi-do
  - Kyunggi-Do
  - Seoul
- Ukraine (6):
  - Dnipro
  - Hlevakha
  - Kharkiv
  - Kiev
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Gopal S, Lane R, Nuamah I, Copenhaver M, Singh J, Hough D, Bach M, Savitz A. Evaluation of Potentially Prolactin-Related Adverse Events and Sexual Maturation in Adolescents with Schizophrenia Treated with Paliperidone Extended-Release (ER) for 2 Years: A Post Hoc Analysis of an Open-Label Multicenter Study. CNS Drugs. 2017 Sep;31(9):797-808. doi: 10.1007/s40263-017-0437-9. PMID 28660406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the long-term (2 year) safety and tolerability of paliperidone extended release (ER) in adolescent patients with schizophrenia. This study was conducted from 27 June 2007 to 18 July 2012 at 55 centers in 10 countries. A total of 400 patients received at least 1 dose of the study drug and were included in the safety analysis.
Pre-assignment Details: Patients enrolled in this study came from 3 different sources: patients who enrolled directly, patients who were randomly assigned to placebo in the R076477PSZ3001 (NCT00518323) study, and patients who were randomly assigned to paliperidone ER in the R076477PSZ3001 (NCT00518323) study.
Groups:
- Placebo/Paliperidone: Patients in this group were previously assigned to placebo in the R076477PSZ3001 (NCT00518323) study. They started with an oral dose of 6 mg tablets daily, regardless of prior treatment assignment in R076477PSZ3001 (NCT00518323). The initial 6 mg daily dose was increased in increments of 3 mg, not more frequently than once every 5 days until the maximum dose of 12 mg daily was reached. If 12 mg was not well tolerated, then the dose could be reduced down to 9 mg daily. Alternatively the dose could be decreased to 3 mg or 1.5 mg daily, if the initial 6 mg dose was not well tolerated.
- Paliperidone (Double-blind)/Paliperidone: Patients in this group were previously assigned to paliperidone extended-release in the R076477PSZ3001 (NCT00518323) study. They started with an oral dose of 6 mg tablets daily, regardless of prior treatment assignment in R076477PSZ3001 (NCT00518323). The initial 6 mg daily dose was increased in increments of 3 mg, not more frequently than once every 5 days until the maximum dose of 12 mg daily was reached. If 12 mg was not well tolerated, then the dose could be reduced down to 9 mg daily. Alternatively the dose could be decreased to 3 mg or 1.5 mg daily, if the initial 6 mg dose was not well tolerated.
- Paliperidone (No Double-blind)/Paliperidone: Patients in this group were directly enrolled into the study and started with an oral dose of 6 mg tablets daily. The initial 6 mg daily dose was increased in increments of 3 mg, not more frequently than once every 5 days until the maximum dose of 12 mg daily was reached. If 12 mg was not well tolerated, then the dose could be reduced down to 9 mg daily. Alternatively the dose could be decreased to 3 mg or 1.5 mg daily, if the initial 6 mg dose was not well tolerated.
Period: Overall Study
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone
Started | 39 | 118 | 243
Completed | 24 | 75 | 121
Not Completed | 15 | 43 | 122
Not completed — Adverse Event | 1 | 2 | 23
Not completed — Lack of Efficacy | 6 | 12 | 27
Not completed — Lost to Follow-up | 3 | 5 | 16
Not completed — Withdrawal by Subject | 5 | 20 | 44
Not completed — Other reasons for withdrawal | 0 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 118 | 243 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 118 | 243 | 400
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.48) | 15.3 (1.59) | 15.3 (1.53) | 15.4 (1.55)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 44 | 92 | 157
  Male | 18 | 74 | 151 | 243
Region of Enrollment [Number; unit: participants]
  Bulgaria | 0 | 0 | 6 | 6
  Estonia | 0 | 0 | 3 | 3
  Finland | 0 | 0 | 3 | 3
  India | 6 | 23 | 35 | 64
  Korea | 0 | 0 | 40 | 40
  Poland | 0 | 0 | 47 | 47
  Romania | 2 | 8 | 10 | 20
  Russia | 18 | 51 | 40 | 109
  Ukraine | 8 | 22 | 18 | 48
  United States of America | 5 | 14 | 41 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experienced Adverse Events as a Measure of Safety and Tolerability
Description: A serious adverse event as defined by the International Conference on Harmonisation (ICH) is any untoward medical occurrence that at any dose results in death, is life-threatening (the subject was at risk of death at the time of the even; it does not refer to an event that hypothetically might have caused death if it were more severe), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to 2 years
Population: The safety analysis set was used for the safety analyses and included all enrolled participants who received at least 1 dose of the open-label study drug as recorded on the electronic case report form. This population was considered as evaluable participants.
Measure: Number; unit: Number of Participants
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 118 | 243 | 400
Number of Participants
  Treatment Emergent Adverse Events (TEAEs) | 32 | 88 | 221 | 341
  Possibly-related TEAEs | 24 | 61 | 185 | 270
  One or More Serious TEAEs | 9 | 4 | 46 | 59

2. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Scores - Last Observation Carried Forward
Description: The PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: The open-label intent-to-treat analysis set was used for the efficacy analyses. All enrolled participants who received at least 1 dose of open-label study drug and had both the baseline and at least 1 postbaseline assessment in the open-label phase were included in this analysis set.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 117 | 237 | 393
Scores on a scale | -18.9 (21.47) | -12.6 (19.92) | -22.4 (22.25) | -19.1 (21.89)

3. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Based on Marder Factors - Last Observation Carried Forward
Description: Neuropsychiatric symptoms of schizophrenia were assessed using the 30-item PANSS scale. PANSS scale provides a total score (sum of scores of all 30 items) and scores for 3 subscales, ie, positive (7 items), negative (7 items), and general psychopathology (16 items) subscales. Each item is scored on a scale of 1 (absent) to 7 (extreme). Positive Factor Score (range: 8 to 56): sum of select scores from positive, negative, and general psychopathology subscales. Negative Factor Score (range: 7 to 49): sum of select scores from negative and general psychopathology subscales. Disorganized Thoughts Factor Score (range: 7 to 49): sum of select scores from positive, negative, and general psychopathology subscales. Uncontrolled Hostility/Excitement Factor Score (range: 4 to 28): sum of select scores from positive and general psychopathology subscales. Anxiety/Depression Factor Score (range: 4 to 28): sum of select scores from general psychopathology subscale. Higher scores indicate worsening.
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: The open label intent-to-treat analysis set was used for the efficacy analyses. All enrolled participants who received at least 1 dose of open label study drug and had both the baseline and at least 1 postbaseline assessment in the open label phase were included in this analysis set.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 117 | 237 | 393
Scores on a scale
  Positive Symptoms | -5.1 (6.45) | -3.4 (6.11) | -7.0 (7.12) | -5.7 (6.94)
  Negative Symptoms | -4.3 (6.30) | -3.8 (4.80) | -5.7 (6.68) | -5.0 (6.18)
  Disorganized Thoughts | -4.8 (5.57) | -3.3 (4.41) | -4.9 (5.52) | -4.4 (5.25)
  Uncontrolled Hostility/Excitement | -2.6 (4.17) | -1.2 (4.41) | -2.1 (4.68) | -1.9 (4.56)
  Anxiety/Depression | -2.1 (3.35) | -0.9 (3.41) | -2.8 (3.61) | -2.2 (3.62)

4. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in the Clinical Global Impression Severity (CGI-S) Scale - Last Observation Carried Forward
Description: The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 117 | 237 | 393
Scores on a scale | -1.0 [-3 to 2] | -1.0 [-3 to 3] | -1.0 [-5 to 3] | -1.0 [-5 to 3]

5. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in the Children's Global Assessment Scale (CGAS) - Last Observation Carried Forward
Description: The CGAS is a 100 point rating scale which measures the psychological, social, and school functioning for children 6 to 17 years of age. The score ranges from 1 to 100, divided into 10 equal intervals to rate the impairment level of general functioning (poor to superior functioning). Higher scores denote better functioning.
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 39 | 117 | 237 | 393
Scores on a scale | 11.3 (16.65) | 8.7 (16.02) | 15.6 (17.77) | 13.1 (17.39)

6. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Motor Speed Domain Test Variable, Finger Tapping Dominant- and Non-Dominant Hand, Scaled - Last Observation Carried Forward
Description: A comprehensive neuropsychological examination that measures different domains of cognitive functioning is provided. They are either assessed as T-scores [mean=50, SD=10 range 1-100]; z-scores [mean=0, SD=1, and can be positive or negative] or scaled scores [mean=10, SD=3, and can be positive or negative]. The theory-of-mind total score is a raw score that ranges from 1 to 100. Higher scores for all scales denote better performance.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 29 | 88 | 154 | 271
Scores on a scale
  Finger Tapping Dominant Hand | 0.2 (1.15) | 0.1 (1.65) | 0.3 (1.36) | 0.2 (1.44)
  Finger Tapping Non Dominant Hand | 0.2 (1.20) | 0.4 (2.05) | 0.2 (1.55) | 0.3 (1.69)

7. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Attention/Working Memory Domain Test Variable Coding, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 27 | 90 | 143 | 260
Scores on a scale | 1.9 (3.25) | 1.5 (2.54) | 0.1 (2.60) | 0.8 (2.75)

8. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Attention/Working Memory Domain Test Variable Digit Span, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 28 | 95 | 159 | 282
Scores on a scale | 0.9 (2.42) | 0.8 (2.81) | 0.8 (2.71) | 0.8 (2.71)

9. Secondary Outcome: Change From Open-label Baseline to Open-label - Cognitive Domain: Verbal Learning and Memory Domain Test Variable Wide Range Assessment of Memory and Learning Story - Total, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 1 | 9 | 17 | 27
Scores on a scale | 0 (NA) — Number of participants analyzed is 1 | 0.6 (3.57) | 1.7 (1.36) | 1.3 (2.33)

10. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Verbal Learning and Memory Domain Test Variable California Verbal Learning Test-Total Trials, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 1 | 11 | 18 | 30
Scores on a scale | 29.0 (NA) — Number of participants analyzed is 1 | 3.5 (12.29) | 8.2 (12.19) | 7.2 (12.70)

11. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Visual Learning and Memory Domain Test Variable, Rey Complex Figure Test - Total, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 29 | 92 | 150 | 271
Scores on a scale | -0.5 (1.56) | -0.3 (2.02) | 0.3 (2.39) | 0.0 (2.21)

12. Secondary Outcome: Change From Open Label Baseline to Open Label Endpoint - Cognitive Domain: Social Cognition Domain Test Variable - Theory of Mind-Total - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 29 | 91 | 149 | 269
Scores on a scale | 3.4 (7.04) | 4.1 (6.68) | 5.6 (9.20) | 4.9 (8.23)

13. Secondary Outcome: Change From Open Label Baseline to Open Label Endpoint - Cognitive Domain: Speed of Processing Domain Test Variable Trials Part A Time: Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 2 | 15 | 21 | 38
Scores on a scale | 1.8 (1.06) | -2.3 (4.97) | 1.5 (7.66) | 0.0 (6.69)

14. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Speed of Processing Domain Test Variable Child Color Trials Test 1 Time: Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 21 | 58 | 101 | 180
Scores on a scale | 0.0 (20.82) | 3.6 (11.90) | 6.2 (14.41) | 4.7 (14.62)

15. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Speed of Processing Domain Test Variable Phonetic Verbal Fluency: Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 21 | 78 | 79 | 178
Scores on a scale | 0.3 (1.48) | 0.2 (1.07) | 0.5 (1.09) | 0.4 (1.14)

16. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Speed of Processing Domain Test Variable Semantic Verbal Fluency, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 20 | 76 | 78 | 174
Scores on a scale | 0.2 (1.23) | 0.1 (0.82) | 0.2 (0.90) | 0.2 (0.91)

17. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Executive Functioning (Reasoning and Problem Solving) Domain Test Variable, Trials Part B Time, Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 0 | 15 | 18 | 33
Scores on a scale |  | 0.2 (2.67) | 0.7 (2.53) | 0.5 (2.57)

18. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint - Cognitive Domain: Executive Functioning (Reasoning and Problem Solving) Domain Test Variable - Wisconsin Card Sort Test-Total Errors: Scaled - Last Observation Carried Forward
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 15 | 66 | 109 | 190
Scores on a scale | 4.3 (11.13) | 4.6 (11.09) | 7.0 (13.16) | 5.9 (12.32)

19. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in the Sleep Visual Analog Scale (VAS): Quality of Sleep - Last Observation Carried Forward
Description: Sleep VAS is a self administered scale that rates the quality of sleep and daytime drowsiness. Participants make a mark on a line to represent how well they have slept in the previous 7 days ("very badly" to "very well") and how often they have felt drowsy within the previous 7 days ("not at all" to "all the time"). The score for each item ranges from 0 to 100 mm. For quality of sleep, a score of 0 indicates "Very badly" and a score of 100 indicates "Very well." For daytime drowsiness, a score of 0 indicates "Not at all" and a score of 100 indicates "All the time." Improvement of the condition is indicated by the positive change for the quality of sleep and the negative change for the daytime drowsiness.
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 36 | 116 | 223 | 375
Scores on a scale | 8.2 (30.51) | 2.7 (18.48) | 9.8 (32.47) | 7.4 (28.78)

20. Secondary Outcome: Change From Open-label Baseline to Open-label Endpoint in the Sleep Visual Analog Scale (VAS): Daytime Drowsiness - Last Observation Carried Forward
Description: as for outcome 19
Time Frame: Baseline, Week 104 or the last post-baseline assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone | Total
Number analyzed (Participants) | 36 | 116 | 223 | 375
Scores on a scale | -7.4 (18.83) | -5.1 (22.39) | -3.9 (32.30) | -4.6 (28.42)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Placebo/Paliperidone | Paliperidone (Double-blind)/Paliperidone | Paliperidone (No Double-blind)/Paliperidone
Serious Adverse Events (participants affected / at risk) | 9/39 | 4/118 | 46/243
Other Adverse Events (participants affected / at risk) | 26/39 | 74/118 | 192/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Paliperidone (N=39) | Paliperidone (Double-blind)/Paliperidone (N=118) | Paliperidone (No Double-blind)/Paliperidone (N=243)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Irritability (General disorders) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Frostbite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 2
Hypokinesia (Nervous system disorders) | 0 | 0 | 1
Oromandibular Dystonia (Nervous system disorders) | 0 | 0 | 1
Speech Disorder (Nervous system disorders) | 0 | 0 | 1
Adjustment Disorder (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 3
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 3
Delusion (Psychiatric disorders) | 0 | 0 | 2
Delusion of Grandeur (Psychiatric disorders) | 0 | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Depressive Symptom (Psychiatric disorders) | 0 | 0 | 1
Flight of Ideas (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 2
Hallucination, Auditory (Psychiatric disorders) | 0 | 0 | 2
Intentional Self-Injury (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Oppositional Defiant Disorder (Psychiatric disorders) | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 2
Schizophrenia (Psychiatric disorders) | 7 | 2 | 21
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 | 0 | 2
Schizophrenia, Undifferentiated Type (Psychiatric disorders) | 0 | 0 | 1
Self Injurious Behaviour (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 7
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 3
Tension (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Paliperidone (N=39) | Paliperidone (Double-blind)/Paliperidone (N=118) | Paliperidone (No Double-blind)/Paliperidone (N=243)
Palpitations (Cardiac disorders) | 2 | 1 | 3
Tachycardia (Cardiac disorders) | 2 | 1 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 14
Nausea (Gastrointestinal disorders) | 1 | 3 | 27
Salivary Hypersecretion (Gastrointestinal disorders) | 2 | 9 | 22
Vomiting (Gastrointestinal disorders) | 0 | 3 | 22
Asthenia (General disorders) | 3 | 3 | 3
Bronchitis (Infections and infestations) | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 18 | 32
Rhinitis (Infections and infestations) | 2 | 2 | 9
Weight Increased (Investigations) | 2 | 12 | 59
Increased Appetite (Metabolism and nutrition disorders) | 2 | 3 | 9
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 1 | 6 | 19
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 14
Akathisia (Nervous system disorders) | 0 | 10 | 42
Dizziness (Nervous system disorders) | 4 | 8 | 13
Dystonia (Nervous system disorders) | 1 | 6 | 13
Headache (Nervous system disorders) | 4 | 9 | 46
Sedation (Nervous system disorders) | 1 | 0 | 14
Somnolence (Nervous system disorders) | 10 | 18 | 45
Tremor (Nervous system disorders) | 1 | 12 | 31
Anxiety (Psychiatric disorders) | 4 | 7 | 14
Insomnia (Psychiatric disorders) | 7 | 11 | 40
Schizophrenia (Psychiatric disorders) | 2 | 10 | 14
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 30
Galactorrhoea (Reproductive system and breast disorders) | 3 | 4 | 9
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.